CLINICAL TRIAL: NCT02246478
Title: A Phase I Study of Single and Multiple Doses of TAS-205 in Patients With Duchenne Muscular Dystrophy
Brief Title: A Study of TAS-205 for Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Taiho10053030
Record Dates: First submitted 2014-09-09; First posted 2014-09-22 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — TAS-205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TAS-205 low dose (Active Comparator)
  Interventions: Drug: TAS-205
- TAS-205 middle dose (Active Comparator)
  Interventions: Drug: TAS-205
- TAS-205 high dose (Active Comparator)
  Interventions: Drug: TAS-205

INTERVENTIONS:
Drug: TAS-205 — * Single-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step, single oral administration after meals
  * Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
  Arms: TAS-205 high dose; TAS-205 low dose; TAS-205 middle dose
Drug: Placebo — * Single-dose phase: 3steps (low dose, middle dose or high dose group), 2 patients/step, single oral administration after meals
  * Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 2 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and pharmacokinetic of TAS-205 in patients with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common fatal genetic disorder diagnosed in childhood, affecting approximately 1 in every 3500 lives male births. DMD patients suffer from a relentless decline in muscle strength that impairs the ability of walking and breathing, resulting in their lives with wheelchairs and loss of upper body function. The objective of this study is to evaluate the safety and pharmacokinetic of TAS-205 after single and multiple doses in DMD patients. It is also evaluated if TAS-205 affects the urinary excretion of pharmacodynamic (PD) marker in DMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to give an informed consent. If applicable, able to give an informed assent.
* Male and >= 5 years and < 16 years of age.
* Bodyweight of >= 15.0 kg and < 75.0 kg.
* Phenotypic evidence of DMD.
* Able to take tablets.
* If taking oral glucocorticosteroids no significant change in total daily dosage or dosing regimen after enrollment.
* Confirmed the urinary PD marker over its criteria.
* Able to follow the study protocol.

Exclusion Criteria:

* Current diagnosis or history of any drug allergy.
* A forced vital capacity (FVC) < 50% of predicted value.
* A left ventricular ejection fraction (EF) < 50% or fractional shortening (FS) < 25% based on echocardiogram (ECHO).
* Ongoing immunosuppressive therapy (other than corticosteroids).
* With severe disease such as hepatic disease, kidney disease and others.
* With any systemic allergic disease or any chronic inflammatory disease.
* Treated with any other investigational agents within 90 days.
* Positive reaction in hepatitis B surface antigen (HbsAg), hepatitis C antibody test (HCV), or human immunodeficiency virus (HIV) test.

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co.,Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- National Center of Neurology and Psychiatry, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants in 21 participants of Single-dose phase discontinued after Single-dose phase. So, 19 participants moved to Multiple-dose phase. And new two participants enrolled in Multiple-dose phase.
Groups:
- Placebo: Placebo: ・Single-dose phase: 3steps (low dose, middle dose or high dose group), 2 patients/step, single oral administration after meals
  ・Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 2 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
- TAS-205 Low Dose; TAS-205 Middle Dose; TAS-205 High Dose: TAS-205: ・Single-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step, single oral administration after meals
  ・Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
Period: Single-dose Phase
Arm/Group | Placebo | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Started | 6 | 5 | 5 | 5
Completed | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Multiple-dose Phase
Arm/Group | Placebo | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Started | 6 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 4
Not Completed | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two participant were discontinued in Single-dose phase, and other two participants were added in Multiple-dose phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 5 | 6 | 23
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 5 | 6 | 23
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 6 | 5 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Source Vocabulary Name for Table Default: CTCAE (4.03)
Time Frame: From the first administration day to the end of the observation period (ie. single-dose phase: 8 days, multiple-doses phase: 14 days)
Population: About repeated-dose period, one participants of placebo group and one of TAS-205 high dose group were excluded from analysis population, due to significant deviation from the protocol.
Measure: Number; unit: participants
Arm/Group | Placebo | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Number analyzed (Participants) | 6 | 6 | 5 | 6
participants
  Single-dose Period | 0 | 3 | 1 | 1
  Repeated-dose Period: number analyzed (Participants) | 5 | 5 | 5 | 4
  Repeated-dose Period | 0 | 1 | 3 | 1

2. Secondary Outcome: Peak Plasma Concentration (Cmax) of TAS-205
Description: Due to inspection missing, some data were not analyzed.
Time Frame: Single-dose phase: immediately before dosing, 0, 0.5, 1, 2, 4, 8, 24, 48 hours post-dose, Multiple-dose phase: Days 1 and 7, immediately before morning dose, 0.5, 1, 2, 4, and 8 hours post-dose and Day 4, immediately before morning dose.
Population: About repeated-dose period, one participants of TAS-205 high dose group was excluded from analysis population, due to significant deviation from the protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Number analyzed (Participants) | 5 | 5 | 5
ng/mL
  Single-dose Period | 839 (383) | 1847 (996) | 3202 (1493)
  Repeated-dose Period (Day 1): number analyzed (Participants) | 5 | 5 | 3
  Repeated-dose Period (Day 1) | 1004 (656) | 1894 (691) | 2635 (2813)
  Repeated-dose Period (Day 7): number analyzed (Participants) | 5 | 5 | 3
  Repeated-dose Period (Day 7) | 891 (297) | 2322 (776) | 4660 (3671)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of TAS-205
Description: Due to inspection missing, some data were not analyzed.
Time Frame: Administration period (ie. single-dose phase: from single administration day to 48 hours after the administration, multiple-dose phase: from the first administration day to 8 hours after the last administration)
Population: About repeated-dose period, one paticipant of TAS-205 high dose group was excluded from analysis population, due to significant deviation from the protocol.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Number analyzed (Participants) | 5 | 5 | 5
ng*hr/mL
  Single-dose Period | 2604 (851) | 5776 (2951) | 9118 (3334)
  Repeated-dose Period (Day 1): number analyzed (Participants) | 5 | 5 | 3
  Repeated-dose Period (Day 1) | 2525 (1208) | 5281 (2553) | 6391 (4731)
  Repeated-dose Period (Day 7): number analyzed (Participants) | 5 | 3 | 5
  Repeated-dose Period (Day 7) | 2642 (673) | 6087 (2561) | 9452 (4405)

4. Secondary Outcome: The Urinary Excretion of PD Marker
Description: Ratio of prostaglandin E2 metabolite / creatinine Due to inspection missing, some data were not analyzed.
Time Frame: Single-dose: Day -1 before administration, 0-24 hr post-dose, and 24-48 hr post-dose, Multiple-doses: Day -1 before administration, 0 hr after administration on Day 1 and 4 to the following day (Day 2 and 5), and 0-24 hr after administration on Day 7.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | TAS-205 Low Dose | TAS-205 Middle Dose | TAS-205 High Dose
Number analyzed (Participants) | 6 | 5 | 5 | 5
ratio
  Single-dose Period | 1.05 (0.14) | 0.92 (0.28) | 1.13 (0.31) | 1.26 (0.46)
  Repeated-dose Period (Day 1): number analyzed (Participants) | 5 | 5 | 5 | 4
  Repeated-dose Period (Day 1) | 1.22 (0.34) | 1.23 (0.33) | 1.07 (0.26) | 1.26 (0.34)
  Repeated-dose Period (Day 7): number analyzed (Participants) | 5 | 5 | 5 | 4
  Repeated-dose Period (Day 7) | 1.22 (0.46) | 1.27 (0.35) | 1.27 (0.21) | 0.76 (0.17)

ADVERSE EVENTS:
Time Frame: From the first administration day to the end of the observation period (ie. single-dose phase: 8 days, multiple-doses phase: 14 days)
Description: Adverse Events were formed by participants of single-dose period and multiple-dose period.
Groups:
- Placebo, Single-dose Phase: Single-dose phase: 3steps (low dose, middle dose or high dose group), 2 patients/step, single oral administration after meals
- TAS-205 Low Dose, Single-dose Phase; TAS-205 Middle Dose, Single-dose Phase; TAS-205 High Dose, Single-dose: Single-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step, single oral administration after meals
- Placebo, Multiple-dose Phase: Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 2 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
- TAS-205 Low Dose, Multiple-dose Phase; TAS-205 Middle Dose, Multiple-dose Phase; TAS-205 High Dose, Multiple-dose Phase: Multiple-dose phase: 3 steps (low dose, middle dose or high dose group), 5 patients/step (the same patients between single- and multiple-dose phases), repeated oral administration for 7 days, BID after meals
Arm/Group | Placebo, Single-dose Phase | TAS-205 Low Dose, Single-dose Phase | TAS-205 Middle Dose, Single-dose Phase | TAS-205 High Dose, Single-dose | Placebo, Multiple-dose Phase | TAS-205 Low Dose, Multiple-dose Phase | TAS-205 Middle Dose, Multiple-dose Phase | TAS-205 High Dose, Multiple-dose Phase
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 3/5 | 1/5 | 1/5 | 0/5 | 1/5 | 3/5 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Single-dose Phase (N=6) | TAS-205 Low Dose, Single-dose Phase (N=5) | TAS-205 Middle Dose, Single-dose Phase (N=5) | TAS-205 High Dose, Single-dose (N=5) | Placebo, Multiple-dose Phase (N=5) | TAS-205 Low Dose, Multiple-dose Phase (N=5) | TAS-205 Middle Dose, Multiple-dose Phase (N=5) | TAS-205 High Dose, Multiple-dose Phase (N=4)
Catheter site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystatin C increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other